CLINICAL TRIAL: NCT03199794
Title: Prospective and Retrospective, Non-interventional Study to Evaluate the Safety and Effectiveness of Obizur in Real-life Practice
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 241501; EUPAS16055 (Registry Identifier: ENCePP)
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Acquired Hemophilia A
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OBIZUR participants: Participants previously treated with OBIZUR and continue to be treated with OBIZUR during the study.
  Interventions: Biological: OBIZUR

INTERVENTIONS:
Biological: OBIZUR — Treating physician will determine treatment regimen and frequency of laboratory and clinical assessments according to routine clinical practice.
  Other Names: Recombinant pFVIII; Porcine Sequence; rpFVIII; Antihemophilic Factor (Recombinant)

SUMMARY:
The study addresses the safety, utilisation and effectiveness of Obizur in the treatment of bleeding episodes in real-life clinical practice in Europe and the United States.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (or legal representative) is willing to provide informed consent
* Participant is being treated or was treated (treatment initiation within 30 days) with Obizur in routine clinical practice

Exclusion Criteria:

* Participant has known anaphylactic reactions to the active substance, hamster protein or to any of the following excipients: Polysorbate 80; sodium chloride; calcium chloride dihydrate; sucrose; Tris Base; Tris HCl; Tri-sodium citrate dihydrate; sterilized water for injections
* Participant has participated in a clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving a medicinal product or device at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A participant with acquired hemophilia (AH) must be prescribed Obizur for the treatment of a bleeding episode by a physician, independent of and prior to the decision to enrol the participant in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Number of AEs and SAEs including seriousness, severity and outcome | From first administration of Obizur up to 180 days after the last administration of Obizur.
  AE - adverse event, SAE - serious adverse event.
Number of AESIs including seriousness, severity, relationship to therapy, outcome, and treatment discontinuation | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Adverse Events of Special Interest (AESI) are as follows: hypersensitivity reactions, thromboembolic events and dose dispensing medication errors.
Number of thromboembolic events | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Thromboembolic events include disseminated intravascular coagulation (DIC), venous thrombosis, pulmonary embolism, myocardial infarction and stroke.
Number of dose dispensing medication errors | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Dose dispensing medication erros include miscalculation of dose while prescribing (calculation of correct dose based on the participant's weight) or administration of the incorrect dose.

SECONDARY OUTCOMES:
Immunogenicity; newly recognized anti-pFVIII inhibitor or increase in titre of anti-pFVIII inhibitors and evolution of titre over time | From first administration of Obizur up to 180 days after the last administration of Obizur.
Obizur treatment regimen, as available | From first administration of Obizur up to 180 days after the last administration of Obizur.
  This may include details of the Obizur treatment regimen utilized, as available
Other medication administered for haemostatic control, as available | From first administration of Obizur up to 180 days after the last administration of Obizur.
  This may include additional medications, treatments and procedures (other than Obizur) undertaken to control a bleeding episode.
Overall effectiveness assessment for resolution of bleeding | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Resolution of bleeding determined as either bleeding stopped or did not stop. If bleeding did not stop, a reason should be provided.
Dose per infusion administered to achieve bleeding control, death or change in haemostatic treatment other than Obizur | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Bleeding control defined as all bleeding stopped.
Number of infusions administered to achieve bleeding control, death or change in haemostatic treatment other than Obizur | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Bleeding control defined as all bleeding stopped.
Time to achieve bleeding control, death or change in haemostatic treatment other than Obizur | From first administration of Obizur up to 180 days after the last administration of Obizur.
  Bleeding control defined as all bleeding stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (26):
- United States (6):
  - University of Florida - Shands, Gainesville, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- AKH - Medizinische Universität Wien, Vienna, Austria
- CHU de Rouen - Hôpital Charles Nicolle, Rouen, France
- Germany (5):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
- Italy (7):
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Universitario Agostino Gemelli, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Rome
  - Istituto Clinico Humanitas, Rozzano
- Radboud University Medical Centre, Nijmegen, Netherlands
- United Kingdom (5):
  - University Hospital Birmingham, Birmingham
  - St James's University Hospital, Leeds
  - Royal Free Hospital, London
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Miesbach W, Curry N, Knobl P, Percy C, Santoro R, Schmaier AH, Trautmann-Grill K, Badejo K, Chen J, Nouri M, Oberai P, Klamroth R. Real-world use of recombinant porcine sequence factor VIII in the treatment of acquired hemophilia A: EU PASS. Ther Adv Hematol. 2024 Sep 2;15:20406207241260332. doi: 10.1177/20406207241260332. eCollection 2024. PMID 39228858
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc64db2bf003ab45d45?idFilter=%5B%22241501